CLINICAL TRIAL: NCT00150332
Title: Linezolid (PNU-10766/PNU10766SS) in the Treatment of MRSA Infections in Patients Whose Conventional Therapy Has Failed, or Who Are Intolerant to Conventional Therapy; an Open-label, Multi-center Trial
Brief Title: Linezolid for the Treatment of Infections Caused by Methicillin Resistant Staphylococcus Aureus in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12600067; A5951054
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Infections, Nosocomial
MeSH Terms: conditions — Cross Infection | interventions — Linezolid

INTERVENTIONS:
Drug: linezolid

SUMMARY:
Use of linezolid in patients with methicillin-resistant Staphylococcus aureus infections in Japan

ELIGIBILITY:
Inclusion Criteria:

* infection due to methicillin-resistant Staphylococcus aureus

Exclusion Criteria:

* hypersensitivity to linezolid

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-01; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Resolution of infection at the time of completion of therapy

SECONDARY OUTCOMES:
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- Japan (16):
  - Pfizer Investigational Site, Kamogawa, Chiba
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Onga-gun, Fukuoka
  - Pfizer Investigational Site, Hiroshima, Hiroshima
  - Pfizer Investigational Site, Sappopro, Hokkaido
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Moriya, Ibaraki
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Kyoto, Kyoto
  - Pfizer Investigational Site, Isahaya, Nagasaki
  - Pfizer Investigational Site, Nagasaki, Nagasaki
  - Pfizer Investigational Site, Kurashiki, Okayama-ken
  - Pfizer Investigational Site, Okayama, Okayama-ken
  - Pfizer Investigational Site, Suita, Osaka
  - Pfizer Investigational Site, Iruma-gun, Saitama
  - Pfizer Investigational Site, Kodaira, Tokyo